CLINICAL TRIAL: NCT05377814
Title: Using Implementation Intentions Plans to Support Public Use of Face Coverings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Chris Keyworth, Lecturer in Psychology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-13300-21577
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Increased Adherence to Wearing Face Coverings

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive control (No Intervention): The (passive) control condition includes the same questionnaire as the experimental group, however participants are not presented with the intervention.
- Intervention (volitional help sheet) (Experimental): Participants in the intervention group will be asked to form implementation intentions with respect to wearing face coverings. Participants will be presented with the stem "If I am tempted not to wear a face covering consistently…" and given 10 options with which to complete as many "if-then" plans as they like. These ten options have been taken from the literature and have been shown to be effective with respect to changing numerous behaviours, including self-harm, smoking, alcohol consumption and physical activity.
  Interventions: Behavioral: Volitional help sheet

INTERVENTIONS:
Behavioral: Volitional help sheet — Participants are asked to choose from a list of strategies for increasing physical activity
  Arms: Intervention (volitional help sheet)

SUMMARY:
The aim of the present research is to test the effectiveness of an implementation intention-based intervention for promoting the wearing of face coverings in three key settings, namely: transport, workplaces and leisure activities.

Each participant will be randomly allocated to one of two conditions. The two conditions are: (1) a control condition, and (2) intervention (form multiple implementation intentions from a drop-down menu). The main outcome measure will be use of face coverings.

DETAILED DESCRIPTION:
Background and study aims

The investigators' previous research showed high levels of adherence to government instructions among a representative sample of the UK adult population during the COVID-19 pandemic (April 2020). The investigators were also able to provide concrete recommendations for interventions to support people's capabilities, opportunities and motivations in order to sustain behaviour change in the long term. One key recommendation was that interventions designed to bolster people's "automatic motivation" (i.e., habits, emotions) would likely lead to the largest improvements in adherence.

However, the research is limited by not looking separately at face coverings, which were not recommended at the time (April 2020), but were made mandatory in certain settings by July 2020. Since July 2020 Government guidance on whether or not people should wear face coverings to protect themselves and others in various settings has fluctuated and is currently (Feb 10 2022) 'recommended'. Vacillations in government advice may undermine future attempts to reinstate mandatory wearing of face coverings, when the need arises.

The investigators' more recent work on the wearing of face coverings specifically, carried out with opportunistic samples of 297 participants from two UK Universities, showed high levels of adherence to face coverings and similarly found that interventions designed to target automatic motivation would similarly have the largest benefits for increasing adherence.

The question then arises as to how one changes automatic motivation at scale in a public health setting. There is a long track record of research showing that implementation intentions are an effective means of changing behaviour, and that such changes in behaviour can be sustained over years. Implementation intentions help people overcome automatic motivation by making the critical situations that may elicit unwanted habits more salient, and ensuring that alternative strategies are deployed. They are best thought of as "if-then" plans: specifying an "if" ensures that triggers to unwanted habits receive greater attention and linking "ifs" with "thens" (e.g., seeking help from someone) ensures that the appropriate responses are automatized and replace the unwanted habit. Forming "if-then" plans thus overcome habits.

Aims

To test the effectiveness of an implementation intention-based intervention for promoting the wearing of face coverings in three key settings, namely: transport, workplaces and leisure activities.

Who can participate?

Adults aged over 18 years of age and have good verbal and written understanding of English

What does the study involve?

Participants complete a series of questionnaires about their wearing of face coverings and are then randomly allocated to one of the two groups. In the intervention group (volitional help sheet), participants will be presented with the stem "If I am tempted not to wear a face covering consistently…" and given 10 options with which to complete as many "if-then" plans as they like. These ten options have been taken from the literature and have been shown to be effective with respect to changing numerous behaviours, including self-harm, smoking, alcohol consumption and physical activity. Participants are asked to make a link (using drop-down menus as part of the online questionnaire) from the situation to their chosen solutions. They can create as many situation and solution pairs as they want. The (passive) control condition includes the same questionnaire as the experimental group (participants are not presented with the intervention). After 6 months participants are asked the same face covering questions to see if the intervention has increased adherence to wearing face coverings.

What are the possible benefits and risks of participating?

By taking part, participants will be helping to understand more about brief interventions to support increased adherence to wearing face coverings. By constructing their own "IF-THEN" plans participants are encouraged to construct their own action plans to deal with potential situations where face coverings would be beneficial.

Below are the main ethical issues and how they will be addressed:

Before giving consent (which will be online, as this is an online-based questionnaire), all project participants will be informed that YouGov will ensure that all data collected is stored confidentially in accordance with their privacy policy.

Participants are still free to withdraw themselves/their data until the data is anonymised (one week after the follow-up questionnaire). There will be no personally identifiable data in the research publication or in the SPSS file that YouGov send to the research team.

Data will not be shared with any researcher or organisation other than in ways detailed on the PIS. Data (which will be anonymised with no identifiable personal information) may be used for secondary analysis within the research team only.

Where is the study run from?

The University of Manchester (UK)

When is the study starting and how long is it expected to run for?

May 2022 to January 2023

Who is funding the study?

This work was supported by funding from the PROTECT COVID-19 National Core Study on transmission and environment, managed by the Health and Safety Executive on behalf of HM Government

Who is the main contact?

1. Prof Christopher J. Armitage Chris.armitage@manchester.ac.uk
2. Dr Chris Keyworth c.keyworth@leeds.ac.uk

Scientific title

Using IF-THEN plans to support public use of face coverings

Study hypothesis

Current study hypothesis as of 14/04/2022:

The condition that completes a volitional help sheet will report higher adherence to wearing of face coverings at follow-up than the control condition

Study design

Two-arm randomised controlled trial

Primary study design

Interventional

Secondary study design

Randomised controlled trial

Trial type

Prevention

Patient information sheet

Not available in web format, please use contact details to request a participant information sheet.

Condition

Increased adherence to wearing face coverings

Intervention

Participants complete a series of questionnaires about their current use of face coverings and are then randomly assigned to one of the two conditions:

1. Participants in the intervention group will additionally be asked to form implementation intentions with respect to wearing face coverings. Participants will be presented with the stem "If I am tempted not to wear a face covering consistently…" and given 10 options with which to complete as many "if-then" plans as they like. These ten options have been taken from the literature and have been shown to be effective with respect to changing numerous behaviours, including self-harm, smoking, alcohol consumption and physical activity.
2. The (passive) control condition includes the same questionnaire as the experimental group (participants are not presented with the intervention).

After 6 months participants are asked to report how often they have worn face coverings to see if the intervention has increased adherence to wearing face coverings.

Intervention type

Behavioural

ELIGIBILITY:
Inclusion Criteria:

Aged 18 and over Good verbal and written understanding of English

Exclusion Criteria:

Aged under 18 years of age Poor verbal and written understanding of English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Use of face coverings | 6 months
  Participants will be asked to rate the extent to which they wear face coverings on 0-100% scales using the items, "Of the time you spent at work / on public transport / doing leisure activities that brought you into contact with other people in indoor spaces (e.g., cinemas, theatres, live music, nightclubs) in the last 7 days, roughly what percentage of it did you spend wearing a face covering?"

SECONDARY OUTCOMES:
Capability, opportunity and motivation (based on Capability, Opportunity, Motivation-Behaviour model) | 6 months
  Measured using the Capability, Opportunity, Motivation questionnaire. Each of the items (0-10 scale) will be analysed separately as these each measure a separate construct. Higher scores indicate higher agreement with statements.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armitage CJ, Keyworth C, Leather JZ, Byrne-Davis L, Epton T. Identifying targets for interventions to support public adherence to government instructions to reduce transmission of SARS-CoV-2. BMC Public Health. 2021 Mar 17;21(1):522. doi: 10.1186/s12889-021-10574-6. PMID 33731056
- [Background] Conroy D, Smith DM, Armitage CJ. Very small effects of an imagery-based randomised trial to promote adherence to wearing face coverings during the COVID-19 pandemic and identification of future intervention targets. Psychol Health. 2023 Sep-Oct;38(10):1288-1308. doi: 10.1080/08870446.2021.2012574. Epub 2022 Jan 11. PMID 35014578
- [Background] Gollwitzer, P. M. (1993). Goal achievement: The role of intentions. European review of social psychology, 4(1), 141-185.
- [Background] Armitage CJ. Evidence that implementation intentions can overcome the effects of smoking habits. Health Psychol. 2016 Sep;35(9):935-43. doi: 10.1037/hea0000344. Epub 2016 Apr 7. PMID 27054302
- [Background] Keyworth C, Epton T, Goldthorpe J, Calam R, Armitage CJ. Acceptability, reliability, and validity of a brief measure of capabilities, opportunities, and motivations ("COM-B"). Br J Health Psychol. 2020 Sep;25(3):474-501. doi: 10.1111/bjhp.12417. Epub 2020 Apr 20. PMID 32314500
- [Derived] Armitage CJ, Keyworth C, Gartland N, Coleman A, Fishwick D, Johnson S, van Tongeren M. Theory-based Trial to Promote Uptake and Sustained Use of Face Coverings During the COVID-19 Pandemic. Ann Behav Med. 2023 Oct 16;57(11):921-928. doi: 10.1093/abm/kaad039. PMID 37656890